CLINICAL TRIAL: NCT04876079
Title: Towards Prevention of Mild-to-moderate Hypoglycemia in Type 1 Diabetes With Oral Glucose at a Higher Blood Glucose Threshold
Brief Title: Prevention of Mild-to-moderate Hypoglycemia in Type 1 Diabetes
Acronym: REVERSIBLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Responsible Party: Principal Investigator, Rémi Rabasa-Lhoret, Full professor, Institut de Recherches Cliniques de Montreal
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2022-1119
Record Dates: First submitted 2021-05-03; First posted 2021-05-06 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Type 1 Diabetes
Keywords: Hypoglycemia; Type 1 diabetes; Carbohydrates
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — Glucose; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 16g of carbohydrates - Plasma glucose < 4.0 mmol/L (Active Comparator): 16g of carbohydrates will be given when glucose levels are below 4.0 mmol/L (management per guidelines)
  Interventions: Other: Test to induce a decline in plasma glucose; Device: Dexcom G6; Other: Dex4; Drug: Insulin
- 16g of carbohydrates - Plasma glucose ≤ 4.5 mmol/L (Active Comparator): 16g of carbohydrates will be given when glucose levels are equal or below 4.5 mmol/L.
  Interventions: Other: Test to induce a decline in plasma glucose; Device: Dexcom G6; Other: Dex4; Drug: Insulin
- 16g of carbohydrates - Plasma glucose ≤ 5.0 mmol/L (Active Comparator): 16g of carbohydrates will be given when glucose levels are equal or below 5.0 mmol/L.
  Interventions: Other: Test to induce a decline in plasma glucose; Device: Dexcom G6; Other: Dex4; Drug: Insulin

INTERVENTIONS:
Other: Test to induce a decline in plasma glucose — Participants will be admitted at the research center at 7:00 after an overnight fast. A venous catheter will be inserted into an arm vein for blood sampling purposes. A subcutaneous insulin bolus will be administered to bring plasma glucose to the glycemic threshold. Oral carbohydrates (16g) will be given when plasma glucose levels are at the target threshold. Sixty minutes after carbohydrates consumption, a standardized meal will be provided and participants will be discharged 90 minutes after the meal.
Device: Dexcom G6 — Participants will have to wear a Dexcom G6 during study interventions
Other: Dex4 — When the glycemic threshold is reach, participants will be given 16g of Dex4
Drug: Insulin — A subcutaneous insulin bolus will be given to induce a decline in plasma glucose and reach the glycemic threshold.

SUMMARY:
According to guidelines, when a mild-to-moderate hypoglycemia occurs (capillary blood glucose < 4.0 mmol/L), 15-20g of rapidly absorbed carbohydrates should be ingested. Patients should re-test and re-ingest 15-20g carbohydrates every 15 minutes until they recover from hypoglycemia. These recommendations were principally based on two studies conducted in the 80s before the introduction of intensive insulin therapy. In practice, only 32-50% of patients follow the current guidelines. In addition, recent studies suggest that under current intensive insulin therapies, an initial correction with 15g of oral glucose may be insufficient to rapidly correct mild-to-moderate hypoglycemia. With the development and increasing usage of newer glucose monitoring technologies, the community is witnessing a shift in hypoglycemia management, from a reactive to a proactive approach (e.g., prevent imminent episodes rather than treating established episodes).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 18 years old
2. Clinical diagnosis of type 1 diabetes for at least one year
3. Treatment with multiple daily insulin injections or insulin pump therapy with insulin analogs (rapid, ultra-rapid and basal insulin)
4. A glycated hemoglobin A1c ≤ 10%

Exclusion Criteria:

1. Clinically significant microvascular complications: nephropathy (eGFR < 40 ml/min), severe proliferative retinopathy as judged by the investigator, neuropathy (particularly diagnosed gastroparesis)
2. Recent (< 3 months) acute macrovascular event (e.g., acute coronary syndrome or cardiac surgery)
3. Known significant cardiac rhythm abnormality based on investigator's judgement
4. Known significant neurological abnormality (e.g., seizure disorder) based on investigator's judgement
5. Ongoing pregnancy or breastfeeding
6. Severe hypoglycemia episode within 1 month of screening
7. Known uncorrected hypokalemia within the past 3 months (potassium < 3.5 mmol/L)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Time spent of glucose levels < 4.0 mmol/L | 60 minutes after carbohydrates consumption

SECONDARY OUTCOMES:
Plasma glucose levels at 5 minutes after carbohydrates consumption | 5 minutes after carbohydrates consumption
Plasma glucose levels at 10 minutes after carbohydrates consumption | 10 minutes after carbohydrates consumption
Plasma glucose levels at 15 minutes after carbohydrates consumption | 15 minutes after carbohydrates consumption
Plasma glucose levels at 20 minutes after carbohydrates consumption | 20 minutes after carbohydrates consumption
Plasma glucose levels at 30 minutes after carbohydrates consumption | 30 minutes after carbohydrates consumption
Plasma glucose levels at 45 minutes after carbohydrates consumption | 45 minutes after carbohydrates consumption
Plasma glucose levels at 60 minutes after carbohydrates consumption | 60 minutes after carbohydrates consumption
Lowest plasma glucose level eached after CHO consumption | 60 minutes after carbohydrates consumption
Time from CHO consumption to the lowest plasma glucose level reached | 60 minutes after carbohydrates consumption
Time from CHO consumption to plasma glucose < 3.5 mmol/L | 60 minutes after carbohydrates consumption
Percentage of participants reaching hypoglycemia (< 4.0 mmol/L) after CHO consumption | 60 minutes after carbohydrates consumption
Percentage of participants for whom hypoglycemia was corrected at 10 minutes after CHO consumption | 10 minutes after carbohydrates consumption
  Only calculated for participants who will have glucose levels < 4.0 mmol/L
Percentage of participants for whom hypoglycemia was corrected at 15 minutes after CHO consumption | 15 minutes after carbohydrates consumption
  Only calculated for participants who will have glucose levels < 4.0 mmol/L
Percentage of participants for whom hypoglycemia was corrected at 20 minutes after CHO consumption | 20 minutes after carbohydrates consumption
  Only calculated for participants who will have glucose levels < 4.0 mmol/L
Percentage of participants for whom hypoglycemia was corrected at 25 minutes after CHO consumption | 25 minutes after carbohydrates consumption
  Only calculated for participants who will have glucose levels < 4.0 mmol/L
Percentage of participants for whom hypoglycemia was corrected at 30 minutes after CHO consumption | 30 minutes after carbohydrates consumption
  Only calculated for participants who will have glucose levels < 4.0 mmol/L
Percentage of participants for whom hypoglycemia was corrected at 35 minutes after CHO consumption | 35 minutes after carbohydrates consumption
  Only calculated for participants who will have glucose levels < 4.0 mmol/L
Percentage of hypoglycemic events that were corrected at 10 minutes after CHO consumption | 10 minutes after carbohydrates consumption
  Only calculated for events with glucose level < 4.0 mmol/L
Percentage of hypoglycemic events that were corrected at 15 minutes after CHO consumption | 15 minutes after carbohydrates consumption
  Only calculated for events with glucose level < 4.0 mmol/L
Percentage of hypoglycemic events that were corrected at 20 minutes after CHO consumption | 20 minutes after carbohydrates consumption
  Only calculated for events with glucose level < 4.0 mmol/L
Percentage of hypoglycemic events that were corrected at 25 minutes after CHO consumption | 25 minutes after carbohydrates consumption
  Only calculated for events with glucose level < 4.0 mmol/L
Percentage of hypoglycemic events that were corrected at 30 minutes after CHO consumption | 30 minutes after carbohydrates consumption
  Only calculated for events with glucose level < 4.0 mmol/L
Percentage of hypoglycemic events that were corrected at 35 minutes after CHO consumption | 35 minutes after carbohydrates consumption
  Only calculated for events with glucose level < 4.0 mmol/L
Percentage of participants requiring a second treatment with carbohydrates at 20 minutes after the first CHO consumption | 20 minutes after carbohydrates consumption
  Only calculated for participants who will have glucose levels < 4.0 mmol/L
Percentage of participants requiring a second treatment with carbohydrates at 40 minutes after the first CHO consumption | 40 minutes after carbohydrates consumption
  Only calculated for participants who will have glucose levels < 4.0 mmol/L
Percentage of participants requiring a second treatment with carbohydrates at 60 minutes after the first CHO consumption | 60 minutes after carbohydrates consumption
  Only calculated for participants who will have glucose levels < 4.0 mmol/L
Percentage of participants experiencing a rebound hyperglycemia (≥ 10.0 mmol/L) within the first hour following the first carbobydrates consumption | 60 minutes after carbohydrates consumption

CONTACTS AND LOCATIONS:
Overall Officials: Rémi Rabasa-Lhoret, Principal Investigator — Institut de recherches cliniques de Montréal
Locations (1):
- Montreal Clinical Research Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No